CLINICAL TRIAL: NCT06085274
Title: Sentinel lympH Node Biopsy With Indocyanine Green in Breast Cancer After NEoadjuvant Chemotherapy (SHINE): A Prospective Clinical Trial
Brief Title: Sentinel lympH Node Biopsy With Indocyanine Green in Breast Cancer After NEoadjuvant Chemotherapy (SHINE)
Acronym: SHINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-6215.0
Record Dates: First submitted 2023-10-01; First posted 2023-10-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Invasive breast cancer; Indocyanine green; Sentinel lymph node biopsy; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG-SLNB (Experimental): This is a prospective within-patient clinical study to assess the accuracy of ICG SLNB compared to standard dual-tracer SLNB in breast cancer patients treated with neoadjuvant chemotherapy. For SLNB, triple localization of the sentinel lymph nodes using blue dye, Tc-99m and ICG will be utilized in each patient.
  Interventions: Procedure: ICG guided sentinel lymph node biopsy

INTERVENTIONS:
Procedure: ICG guided sentinel lymph node biopsy — During sentinel lymph node biopsy the surgeon will inject a volume of 0.1ml divided into 2 doses (0.05ml each) of 2.5mg/mL ICG into the periareolar dermis of the involved breast. Technetium and blue dye will also be administered as per standard of care. The surgeon will assess the axilla with the the SPY-PHI near infrared imaging system to identify and remove ICG-fluorescent nodes; Any other sentinel lymph nodes identified will also be removed as per standard of care. If there is no progression of ICG towards the axilla, or if no ICG sentinel lymph node can be identified, an alternate injection technique involving peritumoural injection at 2-3 locations near the cancer site in the subcutaneous or dermal space of 0.05ml will be utilized.

SUMMARY:
This is a prospective, open-label, within-patient clinical trial to determine the accuracy of Indocyanine green (ICG) guided sentinel lymph node biopsy (SLNB) compared to the standard dual-tracer SLNB in breast cancer patients who have had chemotherapy as a first treatment using a non-inferiority design.

Patients with operable breast cancer treated with chemotherapy and eligible for SLNB will be included in the study. During surgery, ICG will be injected and used to identify fluorescent sentinel nodes using a hand-held imaging camera; radiotracer and blue dye will also be used as per standard protocols. Intraoperative and clinicopathologic outcomes such as complications, characteristics of nodes, false negative rates and feasibility will be assessed. Patients will be asked to complete standardized patient reported outcome questionnaires (Breast-Q, FACT-B+4, VAS) to define the patient experience with this novel technique.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 and ≤ 80
2. Stage I-III core biopsy confirmed invasive breast cancer, who have undergone neoadjuvant chemotherapy and are planned to undergo SLNB with dual tracer (blue dye+Tc-99m)
3. Eastern Cooperative Oncology Group (ECOG) < 2
4. No ICG/iodine allergy
5. Capable of providing informed consent
6. English literacy

Exclusion Criteria:

1. Significant medical comorbidities (ASA 4)
2. Breast cancer stage T4/inflammatory or N2 disease at presentation (SLNB is contra-indicated in this setting)
3. Clinical node positive after neoadjuvant therapy (SLNB is contra-indicated in this setting)
4. Previous axillary surgery or breast/axillary radiotherapy to ipsilateral breast
5. Active pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of ICG SLNB compared to dual-tracer SLNB in post-neoadjuvant chemotherapy treated breast cancer patients. | From Technetium-99 (Tc-99m) injection to the completion of surgery
  Proportion of lymph nodes identified with ICG compared to the proportion of lymph nodes identified with dual tracer (blue dye/Tc-99m gamma probe)

SECONDARY OUTCOMES:
Complications/safety | From time of Technetium-99 (Tc-99m) injection to 30 days after surgery
  Surgical intra-operative and post-operative complications will be collected to determine safety outcomes. All intra-operative complications will be graded using the ClassIntra classification. All post-operative complications (up to 30 days post-surgical treatment) will be graded using the Clavien-Dindo classification. Treatment-related adverse events will be assessed by CTCAE v5.0.
Patient reported outcome measures - Visual Analog Scale | From baseline/enrolment to 12 months from surgery
  Patients' self-report the intensity of their pain. Scale 0-10, where 10 indicated worst pain possible.
Patient reported outcome measures - FACT-B+4 | From baseline/enrolment to 12 months from surgery
  Breast cancer patients' self-report on various dimensions of their Quality of Life: Measures physical well-being (score range 0-28; higher score = worse outcome), social/family well-being (score range 0-28; higher score = better outcome), emotional well-being (score range 0-24; higher score = worse outcome), functional well-being (score range 0-28; higher score = better outcome), breast cancer subscale (score range 0-28; higher score = worse outcome), lymphedema subscale (score range 0-20; higher score = worse outcome).
Patient reported outcome measures - Breast-Q | From baseline/enrolment to 12 months from surgery
  Breast cancer patients' self-report their perceptions of domains of Quality of Life. Scale 0-100; 100 indicates better satisfaction.

OTHER OUTCOMES:
Budget impact analysis | 1 year
  We will quantify all direct costs associated with implementation of ICG guided SLNB in breast cancer and annual operational costs; these will enable a comparison to cost of the current standard SLNB with Tc-99m and blue dye, including nuclear medicine infrastructure, technicians, and additional health care visits.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided